CLINICAL TRIAL: NCT02537886
Title: Development of Patient Centered Virtual Multimedia Interactive Informed Consent Tool to Improve Patient Comprehension and Consent
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1501015262; R21HSO22319-01A1 (Other Grant/Funding Number: AHRQ)
Record Dates: First submitted 2015-08-20; First posted 2015-09-02 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Patient Centered Outcomes Research
Keywords: PCOR

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Evaluation Group: Researchers will conduct a focus group to evaluate VIC after it has been developed and used by patients. Six asthma patients will comprise this post-launch focus group, with the goal of gathering opinions, beliefs, and attitudes about VIC. We will use this information to enhance the generalizability of the VIC approach.
  Interventions: Device: Patient Centered Virtual Multimedia Interactive Informed Consent tool (VIC)

INTERVENTIONS:
Device: Patient Centered Virtual Multimedia Interactive Informed Consent tool (VIC) — Six asthma patients will comprise this post-launch focus group, with the goal of gathering opinions, beliefs, and attitudes about VIC.

SUMMARY:
The Patient Centered Virtual Multimedia Interactive Informed Consent tool (VIC) will be developed as a patient-centered web-based mobile application and will be able to run on mobile devices. The development of VIC is to create a reusable infrastructure for integrating the informed consent process into clinical care and the clinical workflow in a way that enhances patient comprehension while improving the efficiency of obtaining patient consent.

DETAILED DESCRIPTION:
The informed consent process protects patients and ensures ethical conduct of research. For patients to fully understand the content of the informed consent process, it should clearly explain the purpose, process, risks, benefits and alternatives to medical procedures or clinical research as well as a patient's rights and responsibilities. Patient safety and quality of care are at risk if the informed consent process is not delivered in a way that assures patient comprehension.

Adoption of methods that allow researchers to conduct brief and virtual interviews with participants to complete the informed consent process using tablet computers (e.g. iPads) with a comprehensive multimedia library (e.g. video clips, animations, presentations, etc.) to explains the risks, benefits, and alternatives of the clinical care will enhance patient comprehension.

The goal of this project is to help make the conduct of patient centered outcomes research (PCOR) more efficient and more widely implemented by engaging key stakeholders, including patients, through the development and evaluation of a new mobile health (mHealth) informed consent tool to disseminate PCOR findings in informed consent research.

This study will be conducted over a 15 month period and will consist of 6 parts: (1) Front-End Focus Groups, (2) User Requirements Analysis, (3) Screen Prototypes Usability Focus Groups, (4) Design and Implementation, (5) Before Launch Usability Evaluation, (6) After Launch Usability Evaluation. Given the steps in the process and the changing (i.e. different) subjects/participants in each component of the development process, this study registration record primarily summarizes the final step in the development of VIC.

ELIGIBILITY:
Inclusion Criteria:

* Clinician diagnosis of asthma based on National Asthma Education and Prevention Program (NAEPP) guidelines.
* Historical evidence of variable airflow obstruction.
* Subjects are required to speak English.

Exclusion Criteria:

* >10 pack-year smoking history.
* Active smoking within the past year.
* Other chronic lung disease or asthma variant.
* Patients will be excluded if they cannot safely undergo the studies required for participation.
* Patient or clinician refusal to participate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study includes patients from the Yale Center for Asthma and Airway Disease (YCAAD) clinic. Participants for the VIC study will be recruited from the large and diverse asthma population that the YCAAD GenEx 2.0 trial accesses for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06; Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
VIC Focus Group Feedback | 3-5 weeks following the launch of VIC
  Asthma Patients will use the VIC to complete the informed consent on an iPad. Following 3-5 weeks of use, 8-10 users will be selected to take part in a focus group to evaluate the usability of VIC. The intent of this post-launch focus group, will be to gather opinions, beliefs, and attitudes about VIC. The focus group data will be used to arrive at themes that are common among the focus group participants. This feedback will be used to assess the completed VIC tool and inform further development of such tools.

CONTACTS AND LOCATIONS:
Overall Officials: Fuad Abujarad, MD, Principal Investigator — Yale School of Medicine: Dept of Emergency Medicine
Locations (1):
- Yale School of Medicine: Dept of Emergency Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Abujarad F, Peduzzi P, Mun S, Carlson K, Edwards C, Dziura J, Brandt C, Alfano S, Chupp G. Comparing a Multimedia Digital Informed Consent Tool With Traditional Paper-Based Methods: Randomized Controlled Trial. JMIR Form Res. 2021 Oct 19;5(10):e20458. doi: 10.2196/20458. PMID 34665142